CLINICAL TRIAL: NCT04179942
Title: Fractional Exhaled Nitric Oxide and CRP Levels in Egyptian Patients With Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mona abdel mawla Ahmed El wassefy, faculty of medicine Mansoura University, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MS.16.06.82
Record Dates: First submitted 2019-11-19; First posted 2019-11-27 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: OSA
Keywords: FeNO; ;;; Hs-CRP; CPAP; OSA
MeSH Terms: interventions — Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Active Comparator): full night PSG (polysomnogram) was done, fractional exhaled nitric oxide and Hs-CRP were measured
  Interventions: Diagnostic Test: Fractional exhaled nitric oxide and CRP levels
- control (Placebo Comparator): CRP level was measured
  Interventions: Diagnostic Test: Fractional exhaled nitric oxide and CRP levels

INTERVENTIONS:
Diagnostic Test: Fractional exhaled nitric oxide and CRP levels — measurement of FeNO and Hs-CRP after 3months of CPAP

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) was associated with upper and lower respiratory tract inflammation, Fractional exhaled nitric oxide (FeNO) proposed as a marker of airway inflammation, few studies were done on the impact of continuous positive airway pressure (CPAP) on FeNO.

Aim of the work: to study the impact of continued positive airway pressure therapy on exhaled NO and using Hs-CRP as a marker of inflammation in obstructive sleep apnea syndrome.

Patient and Methods: This study is a case-control study including participants were newly diagnosed as OSAS and control recruited from sleep outpatient clinic, full night PSG was done, fractional exhaled nitric oxide and Hs-CRP were measured next morning of PSG, CPAP for moderate to severe OSA patient was advised with measurement of FeNO and Hs-CRP after 3months of CPAP Keywords: FeNO; Hs-CRP; CPAP; OSA. This research did not receive any specific grant from funding agencies in the public, commercial, or not-for-profit sectors.

DETAILED DESCRIPTION:
This study is a prospective 3 months follow up study including only (27) participants as a convenient sample for the cost limitations newly diagnosed as OSA and (10) healthy control.

inclusion characters All participants enrolled in this study

1. were ≥ 18 years old,
2. non-smokers and
3. excluded from any inflammatory disorders (allergy, bronchial asthma, gastro-esophageal reflux disease, cardiovascular diseases, and cerebrovascular diseases) or use of any regular medication including (nasal/inhaled/oral corticosteroids, antihistaminic, cysteinyl leukotriene receptor inhibitors), or
4. had an upper or lower respiratory tract infection 2 weeks prior to sampling. Control healthy subjects were also free from any sleep disorders symptoms. Cases were recruited from Sleep-disordered breathing unit out Patient Clinic in pulmonary medicine department - Mansoura University - Egypt. All participants in this study were evaluated by history taking with stress on OSAS questionnaires, anthropometric parameters measurement and spirometric pulmonary function (FEV1, FVC and FEV1/FVC ) all patients were subjected to laboratory, attended, full-night polysomnography using (SONMOscreenTMplus, SOMNOmedics, (Germany) with AASM standard montage, This included a standardized montage: two-channel electroencephalograms (EEG; C4/A1, C3/A2), bilateral electrooculogram (EOG), submental electromyogram (EMG), bilateral leg EMGs, and electrocardiography (ECG). Airflow was measured using a thermistor (Healthdyne Technologies), the respiratory effort was assessed by inductance plethysmography and oxygen saturation was recorded using a finger probe. The oxygen saturation signal was digitally sampled at 1 Hz and stored both on the PSG record and in a separate monitor for offline analysis.

studies were interpreted according to the last manual scoring criteria. The cases were diagnosed as severe OSA according to the third international classification of sleep disorders. Then they were classified according to apnea-hypopnea index (AHI) into two main groups: cases (AHI ≥5) (n=) and control (AHI˂5) (n=10). Cases were classified into two subgroups into severe OSA (AHI ≥ 30) (n=34) and moderate OSA (AHI (15-30) mild (n=10).

On the next morning of the study 30 min after PSG, the blood sample was collected for measuring of high sensitivity C- reactive protein (HS-CRP) by (The Immunospec Hs-CRP) ELISA, based on the principle of a solid phase enzyme-linked immunosorbent assay [15]. The assay system utilizes a unique monoclonal antibody directed against a distinct antigenic determinant on the CRP molecule.

1. fractional exhaled nitric oxide (FeNO) measurement: was measured by (NO breath®FeNO monitor-Bedfont scientific Ltd) according to international recommendations [16], with a single breath online method at constant flow of 50 mL/s or 12 seconds of exhalation of adults with a sensitivity of one part per billion (ppb) Calibration of the analyzer was automatically performed by the software. Briefly, after inhaling to total lung capacity, the subjects exhaled through a mouthpiece into an exhalation circuit. All subjects were asked to stop eating, drinking, and strenuous exercise for two hours prior to FeNO measurement.
2. CPAP therapy and follow up: 22 of 27 patients with moderate and severe OSA were advised to use CPAP therapy after full-night CPAP titration study in accordance with AASM recommendations [17]Preliminary education and adaptation for CPAP was performed 1hour prior to the beginning of CPAP titration.

   An optimal titration study was defined as one in which an optimal CPAP pressure was reached that normalizes the AHI and eliminates snoring, desaturation, and arousals, and restores a normal flow contour [17] adjusted prescribed CPAP pressure after titration was administered during sleep for at least five hours per night, for at least five days per week for three consecutive months.
3. follow up sessions after CPAP therapy: were adjusted 1,2 and 3 months after starting CPAP therapy for evaluation of patients response and compliance to CPAP, Adherence to the CPAP therapy was evaluated after revision of the download information from the CPAP device.

   Adherence was defined as CPAP use for an average of 4 h on

   ≥ 70% of the nights.
4. (FeNO) was also measured in the three follow up visit with CPAP follow up, however, BMI, spirometric pulmonary function(FEV1, FVC, and FEV1/FVC ) and high sensitivity C- reactive protein (HS-CRP) were measured after 3 months in last follow up visit of the study.

Five patients from 27 were lost in follow up sessions because they did not use CPAP.

Then data were analyzed using SPSS version 16 for Windows® (SPSS Inc, Chicago, IL, USA). Qualitative variables were presented as numbers and percentages. Chi-square test or Fisher exact test of significance was for comparison between groups, as appropriate. Quantitative variables were presented as mean ±SD. They were tested for normality distribution by the Kolmogorov-Smirnov test. In normally distributed variables unpaired t-test (t) was used. In abnormally distributed variables independent Mann-Whitney test (Z) was used. P-value ≤0.05 was considered statistically significant. For the detection of cut off points, we use the receiver operating characteristic (ROC) curve. Sensitivity, Specificity values were used for studying the selected cut off point for validation as a screening tool.

ELIGIBILITY:
Inclusion Criteria:

fractional exhaled nitric oxide and Hs-CRP were measured next morning of PSG, CPAP for moderate to severe OSA patient was advised with measurement of FeNO and Hs-CRP after 3months of CPAP

1. were ≥ 18 years old,
2. non-smokers and
3. excluded from any inflammatory disorders (allergy, bronchial asthma, gastro-esophageal reflux disease, cardiovascular diseases, and cerebrovascular diseases) or use of any regular medication including (nasal/inhaled/oral corticosteroids, antihistaminic, cysteinyl leukotriene receptor inhibitors),
4. or had upper or lower respiratory tract infection 2 weeks prior to sampling.
5. Control healthy subjects were also free from any sleep disorders symptoms. Cases were recruited from Sleep-disordered breathing unit out Patient Clinic in pulmonary medicine department - Mansoura University - Egypt.

Exclusion Criteria:

1. smokers
2. inflammatory disorders
3. cardiovascular disease,
4. on regular medication including (nasal/inhaled/oral corticosteroids, antihistaminic, cysteinyl leukotriene receptor inhibitors) -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Full-night PSG was performed, | one year
  Measurement of FeNO and Hs-CRP with three month intervals of CPAP

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Faculty Chest Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided